CLINICAL TRIAL: NCT01655485
Title: Effect of a Social Script iPAD Application for Children With Autism Spectrum Disorder(ASD) Undergoing Medical Imaging Procedures
Brief Title: Effect of a Social Script iPAD Application for Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Marquette University (Other)
Responsible Party: Principal Investigator, Norah L. Johnson, Assistant Profesor Marquette University, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 255769-1
Record Dates: First submitted 2011-10-11; First posted 2012-08-02 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Anxiety
Keywords: child anxiety; challenging behaviors; time; Parent anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patient teaching (Experimental): ipad application for social script book
  Interventions: Other: Patient teaching

INTERVENTIONS:
Other: Patient teaching — The Social script application is an story book on the iPAD with photos and script explaining the steps of getting a medical image such as a CAT scan from the perspective of the child.
  Other Names: Going to Imaging ipad application

SUMMARY:
The purpose of the research is to test the effectiveness of the social story intervention delivered using the iPAD application "Going to Imaging" on the anxiety, challenging child behaviors, child injuries and completion rates among children with ASD undergoing medical imaging procedures. A secondary purpose is to test the effect of this intervention on the anxiety levels of the parents of ASD children undergoing medical imaging procedures.

Hypotheses:

H1: Children with ASD who are exposed to a story book "Here the investigators go to medical imaging (x-ray)" to prepare for medical imaging compared with children with ASD exposed to treatment as usual (TAU) will have:

1. Lower anxiety as measured by heart rate respiratory rate, and blood pressure (baseline compared to up to two hours later).
2. Exhibit fewer challenging behaviors as measured by a behavior observation scale (developed for the study (up to 2 hours after baseline)
3. Higher procedure completion rate.
4. Shorter time to complete a procedure.
5. Less child injuries.

   H2: Compared to parents of ASD children exposed to treatment as usual (TAU), parents of children with ASD who are exposed to a story book "Here the investigators go to medical imaging (x-ray)" to prepare for medical imaging will have:
6. Lower state anxiety as measured by the State Anxiety Inventory ( baseline ).

DETAILED DESCRIPTION:
Parent state anxiety is measured at baseline with the 20-item State anxiety measure from www.mindgarden.com. Child anxiety is measured at baseline with vital signs (heart rate, blood pressure, respiratory rate). Behaviors will be observed and recorded on the behavior observation tool up to 2 hours after the baseline measure (during the imaging).

ELIGIBILITY:
Inclusion Criteria:

* Children with autism spectrum disorder
* English speaking parent or guardian.

Exclusion Criteria:

* Non-english speaking parent or guardian
* Severe autism as defined by caregiver or health care provider.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2011-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Child behaviors | up to 2 hours
  Child behaviors measured during imaging procedures with the behaviors observation tool created for this study.

SECONDARY OUTCOMES:
Parent anxiety | Baseline
  State anxiety measure www.mindgarden.com

OTHER OUTCOMES:
Child anxiety | Baseline
  Vital signs
Change in parent anxiety | Change from baseline in state anxiety measure to 30 minutes later
  Parent anxiety is measured at baseline www.mindgarden.com and again after the intervention to see if there is a change.
Change in child anxiety | change in child anxiety from baseline to 30 minutes later
  Child anxiety is measured at baseline vital signs and again after the intervention to see if there is a change.

CONTACTS AND LOCATIONS:
Overall Officials: Norah L Johnson, PhD, Principal Investigator — Children's Hospital and Health System Foundation, Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States